CLINICAL TRIAL: NCT06748599
Title: A Comparative Study Between Laser and Manual Removal of Corneal Epithelium for Photorefractive Keratectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sandra Adel Nashed, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: Laser Vs Manual Keratectomy
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Photorefractive Keratectomy
Keywords: removal of corneal epithelium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group A: patients who are assigned for transepithelial PRK
- group B: patients who are mechanical PRK using a spatula

SUMMARY:
Photorefractive keratectomy (PRK) is a laser eye surgery used to ablate the corneal stroma to correct visual refractive errors . PRK was developed in 1983 by Dr. Steven Trokel and colleagues and first performed in 1987 by Dr. Theo Seiler in Berlin. After receiving approval by the US Food and Drug Administration (FDA) in 1996, PRK was briefly the preferred surgical treatment of ametropia as it provided more predictable and stable results than incisional keratotomy. However, the number of PRK procedures fell in the late 1990s with the growing popularity of laser in situ keratomileusis (LASIK).

The study aims to compare the visual and refractive outcomes along with the pain score and patient satisfaction after photorefractive keratectomy in patients who underwent transepithelial or mechanical removal technique

DETAILED DESCRIPTION:
Today, LASIK remains the most commonly performed visual refractive surgery; nonetheless, there remain select situations in which PRK may be preferable, such as post penetrating keratoplasty , in thin corneas , irregular topographies , treatment of some LASIK flap complications or residual refractive errors after LASIK, It is also indicated in patients that have a high risk for traumatic postoperative flap dislocation as athletes .Several modifications of the traditional PRK have been introduced in an attempt to overcome drawbacks of postoperative pain and corneal haze and irregular epithelial healing associated with the procedure .PRK employs an excimer laser ablation of the anterior corneal stroma beneath the epithelium .The first step of PRK is the removal of the superficial epithelial cells, which may be through a variety of techniques such as mechanical removal with spatula , application of a diluted alcohol solution , use a rotatory brush or transepithelial laser . Each of these techniques should be performed quickly to avoid desiccation and skillfully to avoid nicking Bowman's layer.

The first technique, Mechanical debridement, involves using a blunt spatula to scrape off epithelium from the periphery toward the center. The next step is wiping a sponge hydrated with balanced salt solution (BSS) or carboxymethylcellulose 0.5% across the cornea. This technique benefits from not depending on laser optics; however, mechanical debridement tends to be a lengthy process in inexperienced surgeons, which subsequently increases patient anxiety and reduces stromal hydration .

In the late 1990s, Transepithelial PRK was introduced as an alternative laser-assisted method for epithelial removal . The advantages of this method have been cited as minimum surgical time, zero contact of laser machine with corneal surface, shorter time for surface healing and visual correction, and decreased post-operative discomfort and dry eyes,this technique is popular among patients but requires a longer time for mastery.

ELIGIBILITY:
Inclusion Criteria:

* • Age : older than 18 years old .

  * Gender: Include both males and females.
  * Stable refraction for at least 12 months .
  * Intraocular pressure less than 21mmHg.
  * A period without wearing contact lenses (more than 4 days for soft , more than 2 weeks for rigid contact lenses )
  * No history of any Autoimmune disease .
  * The refractive error must be one that can be treated by PRK

Exclusion Criteria:

* _ patients with any eye disease (significant cataract or unstable glaucoma )

  * uncontrolled external disease such as blepharitis, dry eye syndrome, and atopy/allergy.
  * patients with Keratoconus and other abnormalities of the cornea such as corneal ectasias , thinning , edema , interstitial or neurotrophic keratitis and extensive vascularisation .
  * Patients with active systemic connective tissue disease such as systemic lupus erythematosus (SLE) and rheumatoid arthritis (RA)
  * Ineligibility for Surgery: Exclude patients who are not suitable candidates for surgery .
  * Consider excluding pregnant or lactating women .
  * Patients unwilling to participate in the study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the age group between 18 and 45 years will be included in this study. Subjects selected, which will consist of patients with myopia ( less than - 6 D ) will be divided into 2 groups.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 6 month
  best corrected visual acuity (BCVA) will be observed for at least 6 months postoperatively.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edwards JD, Bower KS, Sediq DA, Burka JM, Stutzman RD, Vanroekel CR, Kuzmowych CP, Eaddy JB. Effects of lotrafilcon A and omafilcon A bandage contact lenses on visual outcomes after photorefractive keratectomy. J Cataract Refract Surg. 2008 Aug;34(8):1288-94. doi: 10.1016/j.jcrs.2008.04.024. PMID 18655978
- [Background] Gamaly TO, El Danasoury A, El Maghraby A. A prospective, randomized, contralateral eye comparison of epithelial laser in situ keratomileusis and photorefractive keratectomy in eyes prone to haze. J Refract Surg. 2007 Nov;23(9 Suppl):S1015-20. doi: 10.3928/1081-597X-20071102-07. PMID 18047000
- [Background] Diakonis VF, Pallikaris A, Kymionis GD, Markomanolakis MM. Alterations in endothelial cell density after photorefractive keratectomy with adjuvant mitomycin. Am J Ophthalmol. 2007 Jul;144(1):99-103. doi: 10.1016/j.ajo.2007.03.039. Epub 2007 May 23. PMID 17509511
- [Background] Barreto J Jr, Netto MV, Reis A, Nakano M, Alves MR, Bechara SJ. Topography-guided (NIDEK customized aspheric treatment zone) photorefractive keratectomy with mitomycin C after penetrating keratoplasty for keratoconus: case report. J Refract Surg. 2009 Jan;25(1 Suppl):S131-5. doi: 10.3928/1081597X-20090115-10. PMID 19248542
- [Background] Alio JL, Soria FA, Abbouda A, Pena-Garcia P. Fifteen years follow-up of photorefractive keratectomy up to 10 D of myopia: outcomes and analysis of the refractive regression. Br J Ophthalmol. 2016 May;100(5):626-32. doi: 10.1136/bjophthalmol-2014-306459. Epub 2015 Sep 10. PMID 26359339